CLINICAL TRIAL: NCT04678531
Title: Swabs Containing Tea Tree Oil and Chamomile Oil Versus Baby Shampoo in Patients With Seborrheic Blepharitis: A Double-Blind Randomized Clinical Trial
Brief Title: TTO Swabs Versus Baby Shampoo in Patients With Seborrehic Blepharitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Koç University (Other)
Responsible Party: Principal Investigator, Ceyhun Arici, MD, Associate Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB2021-2
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Seborrheic Blepharitis
Keywords: seborrheic blepharitis; tea tree oil; baby shampoo; swabs; chamomile oil
MeSH Terms: interventions — Chamomile extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Swabs containing tea tree oil and chamomile oil (Experimental): The swabs will be applied on the eyelids twice a day for 8 weeks followed by a discontinuation period of 4 weeks.
  Interventions: Drug: Swabs containing tea tree oil and chamomile oil
- Baby shampoo (Active Comparator): Baby shampoo will be applied on the eyelids twice a day for 8 weeks followed by a discontinuation period of 4 weeks
  Interventions: Drug: Baby shampoo

INTERVENTIONS:
Drug: Swabs containing tea tree oil and chamomile oil — Swabs will be used in 26 patients for 8 weeks and will be discontinued in the following 4 weeks.
  Arms: Swabs containing tea tree oil and chamomile oil
Drug: Baby shampoo — Baby shampoo will be used in 23 patients for 8 weeks and will be discontinued in the following 4 weeks.
  Arms: Baby shampoo

SUMMARY:
The aim of the study was to compare the efficacy of lid swabs containing tea tree oil (TTO) and chamomile oil and baby shampoo (BS) in the treatment of seborrheic blepharitis.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written consent will have a complete ophthalmological examination to determine eligibilty for study entry. At week 0, patients who meet the eligibility requirements will be randomized in a double blind manner (participant and investigator) in a 1:1 ratio using block randomization to lid wipes containing tea tree oil (TTO) and chamomile oil or baby shampoo (twice daily).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of seborrheic blepharitis

Exclusion Criteria:

* Patients with ophthalmological pathologies that may affect the tear film functions including ocular rosacea, contact lens use, history of any ocular surgery, or patients with systemic pathologies or those using systemic medications that may affect the tear film functions
* Patients younger than 18-year-old
* Patients who used any treatment for blepharitis within the 6 months prior to the examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Efficacy of the treatment assessed by the change in Blepharitis Symptom measure (BLISS) score | Change from Baseline at 4 weeks
  BLISS score is calculated according to the answers given to the questionnaire. Higher BLISS scores is related to a worse outcome. (Range is between 0 and 39)
Efficacy of the treatment assessed by the change in Blepharitis Symptom measure (BLISS) score | Change from Baseline at 8 weeks
  BLISS score is calculated according to the answers given to the questionnaire. Higher BLISS scores is related to a worse outcome. (Range is between 0 and 39)
Efficacy of the treatment assessed by the change in Blepharitis Symptom measure (BLISS) score | Change from Baseline at 12 weeks
  BLISS score is calculated according to the answers given to the questionnaire. Higher BLISS scores is related to a worse outcome. (Range is between 0 and 39)

SECONDARY OUTCOMES:
Efficacy of the treatment assessed by the change in Demodex mite count by light microscopy | 0-4-8-12 weeks
  The number of mites in the epilated 4 eyelashes will be counted under microscope.
Efficacy of the treatment assessed by the change in the Schirmer's test results | 0-4-8-12 weeks
  Dry eye evaluation will be made with Schirmer's test.
Efficacy of the treatment assessed by the change in the tear breakup time | 0-4-8-12 weeks
  Dry eye evaluation will be made with tear breakup time.
Efficacy of the treatment assessed by the change in the ocular surface disease index score | 0-4-8-12 weeks
  OSDI scores are calculated according to the responses to the questionnaire. Higher values are related to a worse outcome (range is between 0-100).
Efficacy of the treatment assessed by the change in the non-invasive tear breakup time | 0-4-8-12 weeks
  Dry eye evaluation will be made with non-invasive tear breakup time.
Efficacy of the treatment assessed by the change in the meibomian gland loss | 0-4-8-12 weeks
  Meibomian gland loss will be evaluated using anterior segment analysis system.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided